CLINICAL TRIAL: NCT07125521
Title: Evaluating Medication Adherence of Patients With Gastroesophageal Reflux Disease With Support of the Smartphone Application GERDCare
Acronym: AppGERD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Gastroenterology and Hepatology, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AG2410
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: GERD (Gastroesophageal Reflux Disease)
Keywords: GERD; mobile apps; mobile applications; medication adherence
MeSH Terms: conditions — Gastroesophageal Reflux; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using GERDCare (Experimental): Using the mobile phone application GERDCare (with detailed instructions provided during recruitment)
  Interventions: Other: GERCCare mobile app
- Not using GERDCare (No Intervention): Not using the smartphone application GERDCare

INTERVENTIONS:
Other: GERCCare mobile app — Using the smartphone application GERDCare (with detailed instructions provided during recruitment)
  Arms: Using GERDCare

SUMMARY:
Adherence to GERD treatment, including medication, diet, and lifestyle, is essential for symptom control and complication prevention, yet adherence rates remain low due to various demographic and clinical factors. Digital therapeutics, particularly mobile health applications, have shown promising potential in supporting chronic disease management and improving patient outcomes.

The GERDCare mobile application was developed with direct input from gastrointestinal experts. It is designed to enhance treatment adherence and patient engagement by offering features such as educational resources, symptom tracking, medication reminders, and direct communication between patients and physicians.

The investigators are conducting a single-center, open-label, randomized controlled trial to evaluate the effectiveness of using GERDCare in improving patient adherence. Patients are followed up after four weeks of GERD treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Presents with typical GERD symptoms (regurgitation, heartburn)
* Owns a smartphone and capable of using smartphone applications.

Exclusion Criteria:

* Acute GI conditions (upper GI bleeding, acute peptic ulcer…)
* GI malignancy (esophageal cancer, gastric cancer…)
* Severe chronic comorbidities (heart failure, liver failure, chronic kidney disease…)
* Pregnancy, alcohol abuse, mental health conditions impacting medication adherence or app usage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with good adherence at 4 weeks | 4 weeks after recruitment
  Patients achieved a score of ≥27 points on the Vietnamese Version of the General Medication Adherence Scale (GMAS). Higher scores mean better adherence.

SECONDARY OUTCOMES:
Changes in GERD symptom severity | 4 weeks after recruitment
  GERD symptom severity evaluated by the Gastroesophageal Reflux Disease Questionnaire (GerdQ) Score. The score has a minimum value of 0 and a maximum value of 18. High scores present more severe GERD symptoms. Value ≥ 8 means high probability of GERD.
Proportion of patients with clinical improvement after 4 weeks | 4 weeks after recruitment
  Symptom resolution evaluated clinically
Changes of patients' quality of life after 4 weeks | 4 weeks after recruitment
  Patient's quality of life evaluated by the GERD Quality of Life (GERD-QoL) score. It is an 18-item questionnaire grouped into four subscales (Daily activity, Treatment effect, Diet, and Psychological well-being). The total score was converted to a scale of 0-100, in which 100 means high influence on quality of life caused by GERD symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Gastroenterology and Hepatology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided